CLINICAL TRIAL: NCT01655797
Title: Treating Insomnia in Primary Care: A Study of Effectiveness and Dissemination
Brief Title: Cognitive Behavior Therapy for Insomnia in Primary Care
Acronym: TIRED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala-Örebro Regional Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RFR-10276
Record Dates: First submitted 2012-07-04; First posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Insomnia
Keywords: insomnia; cognitive behavior therapy; primary care
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT (Experimental): The treatment group received manualized CBT-I using a adapted version of a manual designed for use by primary care personnel. Treatment comprised information about sleep and insomnia, methods for medication tapering, sleep hygiene, stimulus control, sleep restriction, progressive muscle relaxation, and dealing with sleep interfering thoughts.
  Interventions: Behavioral: Cognitive behavior therapy for insomnia
- Wait-list (No Intervention): A deferred treatment wait-list condition, with no restrictions placed on the usual care.

INTERVENTIONS:
Behavioral: Cognitive behavior therapy for insomnia — Treatment comprised information about sleep and insomnia, methods for medication tapering, sleep hygiene, stimulus control, sleep restriction, progressive muscle relaxation, and dealing with sleep interfering thoughts.
  Arms: CBT

SUMMARY:
The aim of this study was to investigate the clinical effectiveness of protocol-driven cognitive behavioral therapy (CBT) for insomnia delivered by ordinary primary care personnel (primary care nurses and social workers) in general medical practice with unselected patients, in line with a stepped care approach. The study design was a randomised controlled parallel group design, with allocation to CBT and waiting list control group (WL). Following an active treatment-control period, the control group were re-assigned to CBT. The study hypothesis was that the CBT group would experience less symptoms of insomnia after treatment compared with the WL group. Primary outcome measure was a brief self-report screening form, Insomnia severity index.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled research criteria for chronic insomnia

Exclusion Criteria:

* other untreated sleep disturbance
* pregnancy
* shift work
* concurrent medical or psychiatric condition that could be negatively affected by the treatment
* drug abuse
* severe depression
* dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Insomnia severity index (ISI) | After 9 weeks
  A brief self-report screening form

SECONDARY OUTCOMES:
Change from baseline in sleep-onset latency (SOL) | 9 weeks
  Time to fall asleep, measured with sleep diary
Change from baseline in wake time after sleep onset (WASO) | After 9 weeks
  Time awake during the night, measured with sleep diary
Change from baseline in number of awakenings during the night (NWAK) | After 9 weeks
  Measured with sleep diary
Change from baseline in Sleep efficiency (SE) | After 9 weeks
  Time actually spent sleeping out of the total time in bed (%), measured with sleep diary
Change from baseline in time in bed (TIB) | After 9 weeks
  Measured with sleep diary
Change from baseline in total sleep time (TST) | After 9 weeks
  Measured with sleep diary
Change from baseline in sleep quality (SQ) | After 9 weeks
  Subjective sleep quality (likert scale)
Change from baseline in the fatigue severity scale (FSS) | After 9 weeks
  Self-report questionnaire
Change from baseline in the MOS 36-item short-form health survey, SF-36 | After 9 weeks
  Questionnaire assessing physical and mental health
Change from baseline in the Hospital anxiety and depression scale, HADS | After 9 weeks
  Self-report questionnaire measuring depression and anxiety
Change from baseline in the Epworth sleepiness scale, ESS | After 9 weeks
  Self-report questionnaire assessing daytime sleepiness
Change form baseline in the Pittsburgh sleep quality index (PSQI) | After 9 weeks
  Self-report form assessing sleep quality
Change from baseline in the Minimal insomnia severity scale, MISS | After 9 weeks
  Ultra short screening questionnaire for insomnia
Change from baseline in the Insomnia acceptance questionnaire, IQA | After 9 weeks
  A questionnaire intended to assess acceptance of insomnia
Change from baseline in Body mass index | After 9 weeks
Change from baseline in sagittal abdominal diameter | After 9 weeks
  Abdominal height (cm)
Change from baseline in waist-hip ratio | After 9 weeks
  A ratio of the circumference of the waist to the hips
Change from baseline in blood pressure | After 9 weeks
Change from baseline in heart rate | After 9 weeks
Change from baseline in ALAT | After 9 weeks
  Liver function
Change from baseline in HbA 1c | After 9 weeks
  Glycated hemoglobin
Change from baseline in blood glucose | After 9 weeks
Change from baseline in triglycerides | After 9 weeks
  A type of fat found in the blood
Change from baseline in cholesterol (LDL/HDL) | After 9 weeks
Change from baseline in sleep-onset latency (SOL) | After 18 months
  Time to fall asleep, measured with sleep diary
Change from baseline in wake time after sleep onset (WASO) | After 18 months
  Time awake during the night, measured with sleep diary
Change from baseline in number of awakenings during the night (NWAK) | After 18 months
  Measured with sleep diary
Change from baseline in Sleep efficiency (SE) | After 18 months
  Time actually spent sleeping out of the total time in bed (%), measured with sleep diary
Change from baseline in time in bed (TIB) | After 18 months
  Measured with sleep diary
Change from baseline in total sleep time (TST) | After 18 months
  Measured with sleep diary
Change from baseline in sleep quality (SQ) | After 18 months
  Subjective sleep quality (likert scale)
Change from baseline in the fatigue severity scale (FSS) | After 18 months
  Self-report questionnaire
Change from baseline in the MOS 36-item short-form health survey, SF-36 | After 18 months
  Questionnaire assessing physical and mental health
Change from baseline in the Hospital anxiety and depression scale, HADS | After 18 months
  Self-report questionnaire measuring depression and anxiety
Change from baseline in the Epworth sleepiness scale, ESS | After 18 moths
  Self-report questionnaire assessing daytime sleepiness
Change form baseline in the Pittsburgh sleep quality index (PSQI) | After 18 months
  Self-report form assessing sleep quality
Change from baseline in the Minimal insomnia severity scale, MISS | After 18 months
  Ultra short screening questionnaire for insomnia
Change from baseline in the Insomnia acceptance questionnaire, IQA | After 18 months
  A questionnaire intended to assess acceptance of insomnia
Change from baseline in Body mass index | After 18 months
Change from baseline in sagittal abdominal diameter | After 18 months
  Abdominal height (cm)
Change from baseline in waist-hip ratio | After 18 months
  A ratio of the circumference of the waist to the hips
Change from baseline in blood pressure | After 18 months
Change from baseline in heart rate | After 18 months
Change from baseline in ALAT | After 18 months
  Liver function
Change from baseline in HbA 1c | After 18 months
  Glycated hemoglobin
Change from baseline in blood glucose | After 18 months
Change from baseline in triglycerides | After 18 months
  A type of fat found in the blood
Change from baseline in cholesterol (LDL/HDL) | After 18 months
Change from baseline in the Insomnia severity index (ISI) | After 18 months
  A brief self-report screening form

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Erik Broman, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

REFERENCES:
- [Background] Espie CA, MacMahon KM, Kelly HL, Broomfield NM, Douglas NJ, Engleman HM, McKinstry B, Morin CM, Walker A, Wilson P. Randomized clinical effectiveness trial of nurse-administered small-group cognitive behavior therapy for persistent insomnia in general practice. Sleep. 2007 May;30(5):574-84. doi: 10.1093/sleep/30.5.574. PMID 17552372
- [Derived] Bothelius K, Kyhle K, Espie CA, Broman JE. Manual-guided cognitive-behavioural therapy for insomnia delivered by ordinary primary care personnel in general medical practice: a randomized controlled effectiveness trial. J Sleep Res. 2013 Dec;22(6):688-96. doi: 10.1111/jsr.12067. Epub 2013 Jul 16. PMID 23859625